CLINICAL TRIAL: NCT00481351
Title: Effects of Statin and Ezetimibe Association on Kinetics of Artificial Chilomicrons in Men With Stable Coronary Heart Disease.
Brief Title: Effects of Statin and Ezetimibe Association on Kinetics of Artificial Chilomicrons
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Otavio Celeste Mangili, MD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1068/06
Record Dates: First submitted 2007-05-30; First posted 2007-06-01 (Estimated); Results first posted 2011-01-26 (Estimated); Last update posted 2011-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Coronary Heart Disease
Keywords: artificial chilomicrons kinetics; ezetimibe plus statin; lipid lowering therapy
MeSH Terms: conditions — Coronary Disease | interventions — Simvastatin; Ezetimibe

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- group1 ezetimibe (Experimental): 6 week wash out, followed by 06 week ezetimibe 10mg once a day e then 6 week ezetimibe 10mg plus sinvastatin 20mg for more 6 week.
  Interventions: Drug: Simvastatin 20mg plus ezetimibe 10mg; Drug: ezetimibe
- group 2 simvastatin (Active Comparator): 6 week simvastatin 20mg once a day followed by 6 week simvastatin 80mg once a day.
  Interventions: Drug: simvastatin 20mg; Drug: Simvastatin 80mg

INTERVENTIONS:
Drug: Simvastatin 20mg plus ezetimibe 10mg — simvastatin 20mg plus ezetimibe 10mg once a day for 6 week.
  Arms: group1 ezetimibe
Drug: ezetimibe — ezetimiba 10mg once a day
  Arms: group1 ezetimibe
Drug: simvastatin 20mg — simvastatin 20mg once a day
  Arms: group 2 simvastatin
Drug: Simvastatin 80mg — simvastatin 20mg for 6week and then simvastatin 80mg for the next 6week.
  Arms: group 2 simvastatin

SUMMARY:
Effects of statin and ezetimibe association on kinetics of artificial chylomicrons in men with stable coronary heart disease (CHD).

Background:

The rate (kinetics) of chylomicrons removal from circulation have been correlated with the incidence and severity of atherosclerotic lesions; a number of studies demonstrated lower plasmatic clearance of chylomicrons in patients with CHD compared to patients without this condition. It was also demonstrated a correlation among LDL-C levels and removal of chylomicrons remnants by a technique employing artificial chylomicrons.

The investigators also know that higher doses of more potent statins are more effective in chylomicrons removal than lower doses or less potent statins; nevertheless, the effect of the isolated use of statin has not been completely studied up to now.

Study design:

The investigators propose to study 26 outpatients volunteers with chronic CHD, followed at the Heart Institute - INCOR - of the School of Medicine, University of São Paulo.

Following a period of six weeks of washout from any cholesterol reducer, the kinetics of chylomicrons removal by a technique of emulsion of radiolabeled artificial chylomicrons will be evaluated. Lipid fractions, hepatic enzymes and CK will be measured. Initially patients will be randomly allocated to receive simvastatin 20 mg /day (n= 13) or ezetimibe 10 mg/day (n=13) for six weeks. At the end of this period, kinetics of chylomicrons removal and laboratorial measurements will be repeated (Period 1).

In the next period (Period 2) patients will receive simvastatin 20 mg/ ezetimibe 10 mg (n=13) or simvastatin 80 mg (n=13) for additional six weeks; at the end of this period, the evaluations will be repeated (third and last evaluation).

The aim of this study is to further understand chylomicrons metabolism in patients with chronic coronary disease receiving cholesterol reducers at different dosage regimes.

DETAILED DESCRIPTION:
1-INTRODUCTION:

1.1.Chylomicron metabolism: Chylomicrons are particles formed in the postprandial period and are responsible for transporting blood lipids originating in the diet. These lipoproteins are formed mostly by a core of triglycerides (about 90% of its weight) and small amounts of vitamins and cholesterol esters, surrounded by a phospholipid monolayer. Its protein portion, ie apolipoproteins (apo) remain adhered to the surface of chylomicrons and do not exceed 2% of their total weight, the most common Apo E, CII and CIII, which modulate the activity of lipolytic enzymes or act as ligands for cell receptors.

In the circulation, chylomicrons bind to the endothelial surface of capillaries and triglyceride hydrolysis occurs by the action of lipoprotein lipase (LPL), thereby releasing fatty acids and glycerol to the surrounding cells, thus facilitating their absorption and accumulation in various tissues, especially adipose and muscle. The action of lipase is facilitated by apo CII on the particle surface . This mechanism is extremely important for the transit of energy in the body After this initial phase, the chylomicron remnants, smaller and depleted of triglycerides, are kidnapped in the Disse space and bind to receptors via the hepatic apolipoprotein E. Among these the investigators may mention the very LDL receptors (receptor B / E) and receiver RLP (receptor related protein in LDL). Importantly, apo B48, the main component of chylomicrons and remnants apoprotéico, has only a structural function. Chylomicrons and VLDL share common catabolic pathways regarding LPL and at least in part on the mechanisms of cellular uptake.

Within the classes of lipoproteins, chylomicrons to more rapid removal of plasma, and its half life of about 15 minutes in healthy men. The speed (kinetic) removal of chylomicrons from the circulation has been correlated with the incidence and severity of atherosclerotic injury. Several studies showed lower plasma clearance of chylomicrons in patients with coronary artery disease compared to individuals without atherosclerosis. These findings are found even in normolipemic subjects. Chylomicrons participate in the atherosclerotic process by the generation of foam cells by direct deposition of those remaining in the subendothelial space of arterial wall, and also interference with the reverse transport of colestero. Thus treatments that reduce the plasma concentration of chylomicrons by accelerating its catabolism plasma could be used to prevent atherosclerosis.

Among the methods used to evaluate the plasma kinetics of chylomicron, the investigators bring the lipid emulsion similar to chylomicrons labeled with radioisotopes. They offer an integrated vision and clear steps of the catabolism of chylomicrons in plasma. Several studies have shown that the kinetics of chylomicron is altered in patients with dyslipidemia and / or coronary artery disease (CAD). Defects were found both in lipolysis and the removal of chylomicron remnants, and in CAD patients these process were slowed5. Other studies have also shown that altered kinetics of chylomicrons is a marker of angiographic progression and a more severe course of CAD.

Among the lipid-lowering drugs, statins are the more potent and safe drugs in reducing plasma levels of LDL, leading to decreased LDL cholesterol by 18-55%. They inhibit the hydroxy-methyl-glutaryl coenzyme A reductase (HMGCoA-A reductase), which acts on the synthesis of cholesterol. The enzyme inhibition results in decreased intracellular production of cholesterol by the liver, which leads to increased expression of LDL hepatic receptor, which increases the removal of LDL from the circulation.

The effects of statins on clinical events were studied in several placebo controlled trials randomizing more than 90,000 patients for statin therapy or placebo for 3-5 years time. These studies showed consistently clinical benefit of statins, including reduction of cardiovascular morbidity and mortality, overall mortality, coronary revascularization procedures, and stroke, as demonstrated in a recent meta-analysis. In this group of drugs the investigators find Simvastatin, drug of low cost and high efficacy in reducing cardiovascular events as demonstrated in the study 4S.

Studies have shown that increased expression of LDL receptors in the liver caused by statins leads to increased hepatic uptake of chylomicron artificial emulsions. In this context, it has been demonstrated previously increased plasma removal of chylomicron remnants in patients with coronary disease treated with pravastatin. Likewise, different doses of atorvastatin (10mg and 40mg) were evaluated in relation to intra-vascular metabolism and plasma kinetics of chylomicron emulsion in subjects with dyslipidemia. It was demonstrated that atorvastatin significantly accelerates the removal of chylomicron slowed characteristic of these patients, a dose-dependent, reducing the atherogenic potential of these triglyceride-rich particles in circulation.

Ezetimibe, a new cholesterol absorption inhibitor, emerges as a tool for controlling cholesterol. The drug acts by inhibiting the absorption of dietary cholesterol and bile in the brush border of intestinal epithelium without affecting the absorption of triglycerides and vitamins. Moreover, the glucuronidated ezetimibe undergoes enterohepatic recirculation, repeatedly returning the drug to its site of action. Recent studies suggest that NPC1L1 (Nieman-Pick C1 Like 1 protein) has a critical role in intestinal cholesterol absorption, being established as a direct target for the action ezetimibe18.

Results of several studies in various models have demonstrated the lipid-lowering properties of ezetimibe as monotherapy or in combination with statins. In humans, ezetimibe at a dose of 10mg per day reduces the level of LDL by 12-14%. However, when combined with ezetimibe statins show its therapeutic potential, because its association with low doses of the latter presents lowering effects similar to the use of maximal doses of those statins. Thus the association of low doses of statins with ezetimibe may be an alternative to progressive titration of statin therapy. This would be due to the fact that the association by reducing the concentration of an intense intra-hepatic cholesterol, increase the expression of LDL receptors on the cell membrane of hepatocytes. This fact leads to a higher removal of plasma lipoproteins that bind to these receptors. Recently it was shown that the isolated use of ezetimibe increases the plasma clearance of lipoproteins containing apo B100 (and VLDL remnants and LDL), without however affecting the removal of containing apo B48 (chylomicron remnants). To date, no published study that evaluated the association ezetimibe statin on the kinetics of plasma chylomicrons in research done in medline.

2.RATIONALE: In literature there are already several studies that show that the plasma removal of chylomicron is reduced in subjects with coronary atherosclerosis and that these changes are correlated with greater clinical and angiographic progression of disease.

Therapy with statins in several different schemes proved effective in increasing the kinetics of chylomicron removal in subjects with coronary artery disease, and this effect is dose-dependent. This fact can be explained by the finding that there was an inverse correlation between the plasma clearance of chylomicron remnants and plasma concentrations of LDL-cholesterol. However, to date there is still not clear what the effects of ezetimibe, used alone or in combination with statins, on the chylomicrons. Another aspect to be evaluated is the comparison of titration of statin versus the effects of ezetimibe and statins in their initial doses of chylomicrons, also not previously evaluated

3.METHODS: The study included 30 patients previously diagnosed with stable chronic coronary ischemia in clinical follow-up at the outpatient clinic of the Unit for Chronic Coronary Disease, Heart Institute / INCOR-FMUSP.

After the initial suspension of statin therapy for 6 weeks (washout), patients were randomized into three groups: 12 patients (group 1) treatment with simvastatin 20mg/day, 13 patients (group 2) to therapy with ezetimibe 10mg / day and 5 patients for use of simvastatin 20 mg / day (group 3). In this phase, patients were treated with the drug of choice for 06 weeks and assessed for chylomicron kinetics before and after treatment.

In a second phase, patients received lipid-lowering therapy for optimization of treatment with simvastatin 80 mg / day (group 1) or simvastatin 20 mg / day and ezetimibe 10 mg / day (group 2 and 3) for 6 weeks. Reassessment of the kinetics of chylomicron was held at the end of the second phase.

Data were analyzed kinetics of chylomicrons baseline (without lipid-lowering therapy for a minimum of 6 weeks) after standard-dose monotherapy (first phase) and optimized combination therapy with statins in maximum therapeutic dose or combination of statin and ezetimibe (second phase) in patients with established coronary disease.

Biochemical analysis as well as evaluations of the kinetics of chylomicron were funded by FAPESP No. 0408048-3 entitled "Out of free cholesterol from lipoprotein particles and deposition of cholesterol in the arterial wall: a new mechanism of atherogenesis. The lipid-lowering drugs were supplied by Merck, Sharp & Dohme (simvastatin and ezetimibe).

Regarding the suspension of lipid-lowering drug in patients with stable coronary artery disease (wash-out) for a period of six weeks, there is evidence of no increased risk of acute coronary syndrome in the suspension of statin for up to 6 weeks 24.

The kinetics study of chylomicrons will be carried out as previously published in the literature. The lipid emulsion after preparation shows the following percentage composition: Triolein 76.5 ± 4.1%, free cholesterol 1.9 ± 0.3%, cholesterol ester 11.2 ± 3.0% phospholipids and 10.4 ± 1 3% and sizes ranging from 80 to 100 nm, are made of lipid mixtures emulsified by ultrasonic irradiation and purified by ultracentrifugation in density gradients.

C-cholesteryl oleate and H-Triolina are added (TG, Amershan, UK) mixture for determination of plasma kinetics. The emulsion is then sterilized through a 2μm filter.

Patients are instructed to attend to the laboratory at 8:00 am after fasting for 12 hours to collect blood sample for lipid analysis. The radioactively labeled lipid emulsion is injected as a bolus (volume 200-300μl) containing 74KBp (2μCi) 14C and 148KBp (4μCi) of 3H by antecubital vein catheterization. These concentrations are equivalent to respectively 0.02 and 0.0012 mSv SV radioactive cholesterol and triglycerides. The contralateral antecubital vein is cannulated to obtain blood samples for measurement of radioactivity, saline infusion without heparin infusion was administered slowly to ensure patency of the vein. A saline infusion does not exceed 100ml.

Thereafter, blood samples are collected at predetermined intervals as follows: 2, 4, 6, 10, 15, 20, 30, 45 and 60 minutes after injection of the emulsion.

After collection, blood plasma is separated by centrifugation in 1 ml aliquots, and then transferred to counters containing 7ml of scintillation solution PPO: DM-POPOP: Triton X-100/toluen (5g: 0,5:333 ml/667ml ). The radioactivity in the samples is determined using a Packard 160 TR spectrometer (Packard Meridien, USA).

The estimated time of the metabolism of lipid emulsion is evaluated by compartmental analysis according to the modification of the model proposed by Redgrave and Zench. The delipidation index is then calculated as proposed by Redgrave and Zench, which represents the depletion of the triglyceride content of lipid emulsion before the capture of chylomicrons from the circulation.

The dose of radioactivity even after the three kinetic studies is much lower (0.0636 mSv) maximum annual dose allowed by the International Committee for the Protection of radioactivity 50mSv.

ELIGIBILITY:
Inclusion Criteria:

* Stable coronary heart disease.

Exclusion Criteria:

* Renal and Liver failure
* Hypothyroidism
* Diabetes mellitus
* Neoplasia
* Heart failure.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-06; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raul D. Santos, Physician, Study Director — University of Sao Paulo; Otavio C. Mangili, Physician, Principal Investigator — University of Sao Paulo; Raul C Maranhão, physician, Study Chair — University of Sao Paulo; Ana Carolina M Gagliardi, nutritionist, Study Chair — University of Sao Paulo

REFERENCES:
- [Derived] Mangili OC, Moron Gagliardi AC, Mangili LC, Mesquita CH, Machado Cesar LA, Tanaka A, Schaefer EJ, Maranhao RC, Santos RD. Favorable effects of ezetimibe alone or in association with simvastatin on the removal from plasma of chylomicrons in coronary heart disease subjects. Atherosclerosis. 2014 Mar;233(1):319-25. doi: 10.1016/j.atherosclerosis.2013.12.008. Epub 2014 Jan 17. PMID 24503114

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | group1 Ezetimibe | Group 2 Simvastatin
Started | 13 | 12
Completed | 13 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | group1 Ezetimibe | Group 2 Simvastatin | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 12 | 21
  >=65 years | 4 | 0 | 4
Age Continuous [Mean (Standard Deviation); unit: years] | 61.23 (6.4) | 60.08 (3.42) | 60.68 (4.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 10 | 9 | 19
Waist [Median (Standard Deviation); unit: cm] | 94.85 (9.18) | 97.08 (8.63) | 95.92 (8.81)
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 27.11 (3.41) | 27.96 (3.63) | 27.96 (3.63)
alanine aminotransferase [Mean (Standard Deviation); unit: mg/dl] | 24.23 (11.54) | 20 (4.88) | 22.2 (9.06)
Glucose [Mean (Standard Deviation); unit: mg/dl] | 93.46 (9.40) | 102.17 (11.39) | 97.64 (11.10)
Apolipoprotein A [Mean (Standard Deviation); unit: mg/dl] | 139.18 (29.36) | 136.5 (30.66) | 137.89 (29.39)
Apolipoprotein B [Median (Standard Deviation); unit: mg/dl] | 123.67 (32.99) | 115.74 (19.37) | 119.86 (27.06)
Total cholesterol [Mean (Standard Deviation); unit: mg/dl] | 222.54 (24.35) | 215.33 (33.32) | 219.08 (28.61)
Low Density Lipoprotein [Median (Standard Deviation); unit: mg/dl] | 141.85 (21.91) | 139.42 (22.19) | 140.68 (21.61)
High Density Lipoprotein [Mean (Standard Deviation); unit: mg/dl] | 48.08 (11.88) | 45.08 (13.04) | 46.64 (12.28)
Triglycerides [Mean (Standard Deviation); unit: mg/dl] | 165.23 (80.76) | 213.75 (112.85) | 188.52 (19.60)
cholesteryl ester fractional clearance rate [Mean (Standard Deviation); unit: min-1] | 0.0051 (0.0046) | 0.0046 (0.0029) | 0.0048576 (0.00381)
triglycerides fractional clearance rate [Mean (Standard Deviation); unit: min-1] | 0.0171 (0.0108) | 0.0161 (0.0096) | 0.016602 (0.01004)

OUTCOME MEASURES:

1. Primary Outcome: Cholesteryl Ester Fractional Clearance Rate
Time Frame: 6 weeks
Reporting Status: Not Posted, anticipated posting 2011-07
Measure: Mean (Standard Deviation); unit: min-1

2. Secondary Outcome: Triglyceride Fractional Clearance Rate
Time Frame: 6week
Reporting Status: Not Posted, anticipated posting 2010-11
Measure: Mean (Standard Deviation); unit: min-1

3. Primary Outcome: Low Density Lipoprotein
Time Frame: 12week
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | group1 Ezetimibe | Group 2 Simvastatin
Number analyzed (Participants) | 13 | 12
mg/dl | 74.85 (16.76) | 71.92 (15.35)

4. Secondary Outcome: Alanine Aminotransferase
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | group1 Ezetimibe | Group 2 Simvastatin
Number analyzed (Participants) | 13 | 12
mg/dl | 30.46 (16.08) | 18.33 (8.08)

5. Secondary Outcome: CPK
Time Frame: 12 week
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | group1 Ezetimibe | Group 2 Simvastatin
Number analyzed (Participants) | 13 | 12
mg/dl | 169 (95.41) | 131 (97.54)

6. Secondary Outcome: Total Cholesterol
Time Frame: 12 week
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | group1 Ezetimibe | Group 2 Simvastatin
Number analyzed (Participants) | 13 | 12
mg/dl | 152.61 (26.36) | 148.29 (21.29)

7. Secondary Outcome: High Density Lipoprotein
Time Frame: 12 week
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | group1 Ezetimibe | Group 2 Simvastatin
Number analyzed (Participants) | 13 | 12
mg/dl | 51.31 (16.33) | 44.33 (14.13)

ADVERSE EVENTS:
Arm/Group | group1 Ezetimibe | Group 2 Simvastatin
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/13 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No